CLINICAL TRIAL: NCT01269463
Title: A Randomized, Double-Blind Study of the Time Course of Response to Biphentin® Methylphenidate Hydrochloride ER Capsules Compared to Placebo in Children 6 to 12 Years With Attention Deficit Hyperactivity Disorder in Analog Classroom Setting
Brief Title: Time Course of Response to Methylphenidate HCl ER Capsules in Children 6 to 12 Years With ADHD in Classroom Setting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhodes Pharmaceuticals, L.P. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP-BP-EF001
Record Dates: First submitted 2010-12-31; First posted 2011-01-04 (Estimated); Results first posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Attention Deficit Hyperactivity Disorder; ADHD
Keywords: Attention deficit; Hyperactivity; Impulsivity; Inattention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm; Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: All subjects entered the Open-Label Dose optimization phase and were titrated until an optimized dose of Methylphenidate hydrochloride Extended Release capsule was achieved. Completing subjects then entered the randomized Double-blind Phase (crossover).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open Label Phase Then 2-week Double Blind Phase (Placebo First, Then Methylphenidate HCl ER Capsule) (Experimental): Open Label Phase: Subjects were dose optimized over a 2 to 4 week period. All subjects began at an initial Methylphenidate hydrochloride extended release capsules dose of 15 mg and were titrated weekly to an optimal dose using strengths of 15, 20, 30, up to the maximum of 40 mg/day.
  Double Blind Phase (2-weeks):
  Placebo: Capsule without active drug for 1 week Methylphenidate HCl ER Capsule: An optimized dose of Methylphenidate hydrochloride extended release capsules (15, 20, 30, or 40 mg) for 1 week Dosed once daily in the morning
  Interventions: Drug: Methylphenidate Hydrochloride Extended Release Capsule; Drug: Placebo
- Open Label Phase Then 2-week Double Blind Phase (Methylphenidate HCl ER Capsule First, Then Placebo) (Experimental): Open Label Phase: Subjects were dose optimized over a 2 to 4 week period. All subjects began at an initial Methylphenidate hydrochloride extended release capsules dose of 15 mg and were titrated weekly to an optimal dose using strengths of 15, 20, 30, up to the maximum of 40 mg/day.
  Double Blind Phase (2-weeks):
  Methylphenidate HCl ER Capsule: An optimized dose of Methylphenidate hydrochloride extended release capsules (15, 20, 30, or 40 mg) for 1 week Placebo: Capsule without active drug for 1 week Dosed once daily in the morning
  Interventions: Drug: Methylphenidate Hydrochloride Extended Release Capsule; Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride Extended Release Capsule — An optimized dose of Methylphenidate Hydrochloride Extended Release Capsules 15, 20, 30 or 40 mg to be dosed once daily
  Other Names: Biphentin®
Drug: Placebo — Capsule without active drug
  Other Names: Biphentin placebo

SUMMARY:
The time course of response following one dose of a new methylphenidate hydrochloride extended release capsule is studied in children 6-12 years in a simulated laboratory classroom setting. Biphentin methylphenidate hydrochloride extended release capsule has been formulated for daily dosing to provide treatment of a child with Attention deficit hyperactivity disorder (ADHD) for the substantial day.

DETAILED DESCRIPTION:
Biphentin methylphenidate hydrochloride (HCl) extended release (ER) capsules is provided in multiple strengths of 10, 15, 20, 30, 40, 50, and 60 mg to be administered once daily. Once daily dosing is intended to provide treatment for the substantial day.

For current analog classroom study each eligible subject will be optimized at 15, 20, 30, or 40 mg in a timeframe of five weekly periods. In the sixth week each subject will be randomized double-blind to receive either active comparator at the optimized dose or placebo comparator treatment. The first classroom session will be held at the end of the week, when efficacy measurements including Swanson, Kotkin, Agler, M-Flynn, Pelham Rating Scale (SKAMP) and Permanent Product Measure of Performance (PERMP) tests will be administered. At the beginning of the following week, the subjects will be crossed-over to the corresponding active comparator or placebo comparator treatment. The second classroom session will be held at the end of the second double-blind week, when the same efficacy measurements will be administered.

Various safety and tolerability, and quality of life assessments will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 6 to 12.
2. ADHD diagnosis with ADHD Rating Scale - 4th Edition scores ≥ 90th percentile.
3. In need of treatment for ADHD and able to have 2-day washout from previous medication.
4. Females of child-bearing potential not pregnant and practice birth control.
5. Subject and parent/guardian willing to comply with protocol.
6. Signed consent and assent.

Exclusion Criteria:

1. Estimated Full Scale intellectual level below 80 using Wechsler Abbreviated Scale of Intelligence.
2. Current primary psychiatric diagnosis of: severe anxiety disorder, conduct disorder, psychotic disorders, pervasive developmental disorder, eating disorder, obsessive-compulsive disorder, major depressive disorder, bipolar disorder, substance use disorder, chronic tic disorder, personal or family history of Tourette's Syndrome.
3. Chronic medical illnesses: seizure, hypertension, thyroid disease, cardiac, family history of sudden death, glaucoma.
4. Use of psychotropic CNS meds having effect exceeding 14 days from screening.
5. Planned use of prohibited drugs.
6. Is pregnant or breast-feeding.
7. Significant ECG or laboratory abnormalities.
8. Experimental drug or medical device within 30 days prior to screening.
9. Hypersensitivity to methylphenidate.
10. Inability or unwillingness to comply with protocol.
11. Well controlled on current ADHD treatment.
12. Inability to take oral capsules.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2011-01-19 (Actual); Primary Completion 2011-06-18 (Actual); Study Completion 2013-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-wei Chang, Ph.D., Study Director — NuTec Incorporated; Sharon B. Wigal, Ph.D., Principal Investigator — University of California, Irvine / Child Development Center; Robert Kupper, Ph.D., Study Chair — Rhodes Pharmaceuticals, L.P.
Locations (1):
- University of California, Irvine/Child Development Center, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wigal SB, Greenhill LL, Nordbrock E, Connor DF, Kollins SH, Adjei A, Childress A, Stehli A, Kupper RJ. A randomized placebo-controlled double-blind study evaluating the time course of response to methylphenidate hydrochloride extended-release capsules in children with attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2014 Dec;24(10):562-9. doi: 10.1089/cap.2014.0100. PMID 25470572

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Start Date: 19 January 2011 (First subject screened) Double-Blind Phase Completion Date: 18 June 2011 (Last subject visit in Double-Blind phase) Compassionate Use Phase Completion Date: 13 March 2013 (Last subject visit in Compassionate Use phase)
Pre-assignment Details: Approximately 27 otherwise healthy pediatric subjects (aged 6 to 12) diagnosed with ADHD by DSM-IV-TR™ criteria were planned to participate in the study so that approximately 24 subjects would complete the Double-Blind phase. Subjects were to be randomized into 2 sequences with approximately 12 subjects in each sequence
Period: First Intervention
Arm/Group | Open Label Phase Then 2-week Double Blind Phase (Placebo First, Then Methylphenidate HCl ER Capsule) | Open Label Phase Then 2-week Double Blind Phase (Methylphenidate HCl ER Capsule First, Then Placebo)
Started | 13 | 13
Completed | 11 | 11
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Second Intervention
Arm/Group | Open Label Phase Then 2-week Double Blind Phase (Placebo First, Then Methylphenidate HCl ER Capsule) | Open Label Phase Then 2-week Double Blind Phase (Methylphenidate HCl ER Capsule First, Then Placebo)
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Third Intervention
Arm/Group | Open Label Phase Then 2-week Double Blind Phase (Placebo First, Then Methylphenidate HCl ER Capsule) | Open Label Phase Then 2-week Double Blind Phase (Methylphenidate HCl ER Capsule First, Then Placebo)
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects enrolled in the open-label dose optimization phase and received at least one dose of study drug; 4 subjects withdrew from the study during this phase
Groups:
- Safety Population: All subjects entering open label dose optimization phase (Safety Population) and received at least one dose of study drug
Arm/Group | Safety Population
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.7 (1.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 21
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Comparison Following Treatment Between Drug and Placebo Using Evaluation by SKAMP Combined, Attention, and Deportment Scales
Description: Comparison of Swanson, Kotkin, Alger, M-Flynn and Pelham (SKAMP) Combined, Attention, and Deportment Scales following drug dose versus placebo.
  The SKAMP scale is a validated rating scale that assesses behavioral symptoms of ADHD in a classroom setting using a 7-point impairment scale (0 = none through 6 = maximal impairment). The SKAMP total score comprises 13 items, with individual total scores ranging from 0 to 78 (lower scores mean better outcome). The SKAMP-D subscale evaluates deportment, including interacting with other children, interacting with adults, remaining quiet according to classroom rules, and staying seated according to classroom rules. The SKAMP-A subscale is a measure of attention and evaluates getting started on assignments, sticking with tasks, attending to an activity, and making activity transitions. The SKAMP quality of work subscale includes 3 items: completing assigned work, performing work accurately, and being careful and neat while writing or drawing.
Time Frame: Average over all post-dose time points (1.0, 2.0, 3.0, 4.5, 6.0, 7.5, 9.0, 10.5, and 12 hours)
Population: 20 subjects were in the evaluable population, defined as subjects who completed SKAMP assessments for all the study time points on study days 35 and 42, and who received the scheduled treatment in both periods during the double-blind phase. Two (2) subjects were excluded from the evaluable population due to protocol deviations.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Methylphenidate HCl ER Capsules: Methylphenidate hydrochloride extended release capsules
  Methylphenidate Hydrochloride Extended Release Capsules: Methylphenidate Hydrochloride Extended Release Capsules to be dosed once daily
- Capsule Without Active Drug: Double blind crossover assignment of the placebo comparator.
  Placebo: Capsule without active drug
Arm/Group | Methylphenidate HCl ER Capsules | Capsule Without Active Drug
Number analyzed (Participants) | 20 | 20
units on a scale | 1.46 (0.52) | 2.03 (0.92)
Statistical Analysis 1: Comparison: Methylphenidate HCl ER Capsules vs Capsule Without Active Drug; Test type: Superiority or Other; p < 0.01, ANCOVA

2. Secondary Outcome: Comparison Following Treatment With Drug or Placebo Using PERMP (Permanent Product of Arithmetic) Evaluations
Description: Comparison of PERMP measurement scores following drug dose versus placebo (math-correct).
  The Permanent Product Measure of Performance (PERMP), is a 5-page test consisting of 80 math problems per page (total of 400 problems) and evaluates effortful performance in the classroom as a measure of efficacy. Participants are instructed to work at their seats and to complete as many problems as possible in 10 minutes. The appropriate level of difficulty for each student was determined previously based on results of a math pretest administered at screening. Performance was evaluated using PERMP-A) and PERMP-C scores.
  Measures obtained from these tests include the number of problems attempted (Math-Attempted; PERMP-A) and the number of problems answered correctly (Math-Correct; PERMP-C). Higher scores are better. The responses are reviewed by comparing them to an answer template, and they are triple-checked for accuracy
Time Frame: 12 hours post-dose
Population: 20 subjects were in the evaluable population, defined as subjects who completed PERMP assessments for all the study time points on study days 35 and 42, and who received the scheduled treatment in both periods during the double-blind phase. Two (2) subjects were excluded from the evaluable population due to protocol deviations.
Measure: Least Squares Mean (Standard Deviation); unit: Number of Problems
Arm/Group | Methylphenidate HCl ER Capsules | Capsule Without Active Drug
Number analyzed (Participants) | 20 | 20
Number of Problems
  PERMP-A | 92.85 (48.01) | 80.30 (55.31)
  PERMP-C | 86.85 (49.29) | 74.80 (57.41)
Statistical Analysis 1: Comparison: Methylphenidate HCl ER Capsules vs Capsule Without Active Drug; Test type: Superiority or Other; p < 0.01, ANCOVA

ADVERSE EVENTS:
Time Frame: 11 weeks
Groups:
- Methylphenidate HCl ER During Open Label Phase: Open Label Phase (Period 1): Subjects were dose optimized over a 2 to 4 week period. All subjects began at an initial Methylphenidate hydrochloride extended release capsules dose of 15 mg and were titrated weekly to an optimal dose using strengths of 15, 20, 30, up to the maximum of 40 mg/day.
- Methylphenidate HCl ER Capsules During Double Blind Phase: Double blind crossover assignment of Methylphenidate hydrochloride extended release capsules
  Double Blind Phase (2-week crossover): patients receiving Methylphenidate hydrochloride extended release capsules (15, 20, 30, or 40 mg) for 1 week either on period 2 or period 3 depending on randomization.
  Dosed once daily in the morning
- Capsule Without Active Drug During Double Blind: Double blind crossover assignment of the placebo comparator.
  Double Blind Phase (2-week crossover): patients receiving Placebo for 1 week either on period 2 or period 3 depending on randomization.
  Dosed once daily in the morning
  Placebo: Capsule without active drug
Arm/Group | Methylphenidate HCl ER During Open Label Phase | Methylphenidate HCl ER Capsules During Double Blind Phase | Capsule Without Active Drug During Double Blind
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 23/26 | 7/21 | 3/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate HCl ER During Open Label Phase (N=26) | Methylphenidate HCl ER Capsules During Double Blind Phase (N=21) | Capsule Without Active Drug During Double Blind (N=22)
Emesis (Gastrointestinal disorders) | 3 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 1
Pyrexia (General disorders) | 4 | 2 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Otitis Media (Infections and infestations) | 2 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 6 | 0 | 0
Headache (Nervous system disorders) | 6 | 3 | 0
Insomnia (Nervous system disorders) | 8 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 0 | 0
Emotional Distress (Psychiatric disorders) | 2 | 1 | 0
Irritability (Psychiatric disorders) | 5 | 0 | 1
Mood Swings (Psychiatric disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is restricted from using, disclosing, presenting, or publishing trial information without the prior written consent from the Sponsor